CLINICAL TRIAL: NCT00005324
Title: Genetic and Epidemiologic Studies of Premature Coronary Artery Disease - SCOR in Arteriosclerosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4105; 5P50HL047212-05 (NIH); P50HL027341-15 (NIH); P50HL014237 (NIH); P50HL047151 (NIH); P50HL014197 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To identify genetic mechanisms controlling apolipoprotein levels and other 'non-traditional' risk factors in families ascertained through probands with premature coronary artery disease (CAD).

DETAILED DESCRIPTION:
BACKGROUND:

Preliminary work for this project was carried out as part of the Johns Hopkins Coronary Artery Disease study (R01-HL-34791) which provided extensive data on families ascertained through equal numbers of white male and female probands undergoing elective angiography.

DESIGN NARRATIVE:

The study, a subproject within an Arteriosclerosis SCOR, had three components. In Component 1, the group of 203 probands under study R01HL34791 was expanded with an additional 50 black patients undergoing angiography, meeting identical criteria. In Component 2, segregation analysis was carried out on lipoproteins, apolipoproteins, and selected non-traditional risk factors on families of all probands and the etiologic heterogeneity among different groups of families was tested. In Component 3, linkage was tested between putative Mendelian loci defined in Component 2 and markers in and around candidate loci involved in lipid metabolism. Preliminary results provided evidence of Mendelian control for apolipoprotein A1 and B, and the candidate loci examined included apo B, lipoprotein lipase, and the A1-CIII-A4 gene cluster. The major hypothesis was that these apolipoprotein levels and other non-traditional risk factors might be under genetic control. Genetic analysis of these risk factors was used to direct molecular studies to identify specific mutations.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-01; Study Completion 1996-11 (Actual)

REFERENCES:
- [Background] Mal'tsev VI, Kovalenko VM. [The main trends in the development of a therapeutic service in Ukraine]. Lik Sprava. 1994 Feb;(2):3-9. No abstract available. Ukrainian. PMID 8073714
- [Background] Coresh J, Beaty TH, Prenger VL, Xu J, Kwiterovich PO Jr. Segregation analysis of HDL3-C levels in families of patients undergoing coronary arteriography at an early age. Arterioscler Thromb Vasc Biol. 1995 Sep;15(9):1307-13. doi: 10.1161/01.atv.15.9.1307. PMID 7670942